CLINICAL TRIAL: NCT00113711
Title: Promoting Smoking Cessation and Reducing Weight Gain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 184; R01HL052577 (NIH)
Record Dates: First submitted 2005-06-09; First posted 2005-06-10 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases | interventions — Diet, Reducing

INTERVENTIONS:
Behavioral: smoking cessation
Behavioral: reducing diet

SUMMARY:
To test whether a behavioral intervention could indeed achieve the dual goals of promoting smoking cessation and minimizing weight gain.

DETAILED DESCRIPTION:
BACKGROUND:

When the study began in 1995, more females were initiating cigarette smoking, and a growing proportion cited fear of gaining weight as a major reason for refusing to even attempt quitting smoking. It had not yet been possible, however, to prevent post- cessation weight gain through dieting or behavioral treatment without undermining abstinence from smoking. The investigators proposed that prior interventions had been unsuccessful because: (a) their weight management interventions were too complex; (b) the programs thwarted a need of the patient in nicotine withdrawal to eat hedonically appealing, high-carbohydrate snacks; and (c) the programs heightened patients' emphasis on weight control at the expense of their emphasis on smoking cessation by asking them to initiate weight control before or simultaneously with quitting smoking.

DESIGN NARRATIVE:

The investigators collected pilot data on a promising 16-week intervention that they called the LATE WEIGHT PLAN because it emphasized smoking cessation for the first half of treatment and integrated weight management for the last half. The weight management module included a pre-packaged meal plan; high-carbohydrate, low-fat snacks; and low-intensity aerobic exercise. All patients continued in the weight management phase of treatment, regardless of whether they had succeeded in quitting smoking or were preparing to make new quit attempts. Based on pilot findings, the investigators estimated the point prevalence of smoking cessation for the LATE WEIGHT PLAN group to be 74% at the end of treatment, with weight gain less than 5 lb. An EARLY WEIGHT PLAN group controlled for the timing of the intervention, using the same target quit smoking date and 16 week program but integrating the weight management module into the first 8 weeks of treatment. Like others, they found that EARLY weight management efforts, while they may have prevented weight gain, apparently did so at some cost to smoking cessation, which they estimated to be 42% at 4 months. Finally, a CESSATION ONLY group controlled for the presence of a weight management intervention, by dealing exclusively with smoking cessation for the entire 16 week program. The CESSATION ONLY group had attained the worst outcome in terms of weight control and an intermediate outcome in terms of abstinence at the end of treatment (50%). By randomizing 315 female smokers to the three treatments and comparing abstinence and weight gain after 4 months of treatment and 6 month follow-up (10 months), they tested whether a behavioral intervention could indeed achieve the dual goals of promoting smoking cessation and minimizing weight gain.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
A total of 315 female smokers.

Max Age: 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-01; Study Completion 1999-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Spring — University of Illinois at Chicago

REFERENCES:
- [Background] Persky I, Spring B, Vander Wal JS, Pagoto S, Hedeker D. Adherence across behavioral domains in treatment promoting smoking cessation plus weight control. Health Psychol. 2005 Mar;24(2):153-60. doi: 10.1037/0278-6133.24.2.153. PMID 15755229
- [Background] Sanchez-Johnsen LA, Spring BJ, Sommerfeld BK, Fitzgibbon ML. Weight concerns and smoking in Black and White female smokers. Addict Behav. 2005 Mar;30(3):601-5. doi: 10.1016/j.addbeh.2004.07.007. PMID 15718079
- [Background] Sanchez-Johnsen LA, Fitzgibbon ML, Ahluwalia JS, Spring BJ. Eating pathology among Black and White smokers. Eat Behav. 2005 Feb;6(2):127-36. doi: 10.1016/j.eatbeh.2004.08.011. PMID 15598599
- [Background] Spring B, Pagoto S, Pingitore R, Doran N, Schneider K, Hedeker D. Randomized controlled trial for behavioral smoking and weight control treatment: effect of concurrent versus sequential intervention. J Consult Clin Psychol. 2004 Oct;72(5):785-96. doi: 10.1037/0022-006X.72.5.785. PMID 15482037
- [Background] Doran N, Spring B, McChargue D, Pergadia M, Richmond M. Impulsivity and smoking relapse. Nicotine Tob Res. 2004 Aug;6(4):641-7. doi: 10.1080/14622200410001727939. PMID 15370160
- [Background] Katsutani N, Shionoya H. Drug-specific immune responses induced by procainamide, hydralazine and isoniazid in guinea-pigs. Int J Immunopharmacol. 1992 May;14(4):673-9. doi: 10.1016/0192-0561(92)90130-d. PMID 1521934
- [Background] Cook JW, Spring B, McChargue D, Hedeker D. Hedonic capacity, cigarette craving, and diminished positive mood. Nicotine Tob Res. 2004 Feb;6(1):39-47. doi: 10.1080/14622200310001656849. PMID 14982686
- [Background] Spring B, Pagoto S, McChargue D, Hedeker D, Werth J. Altered reward value of carbohydrate snacks for female smokers withdrawn from nicotine. Pharmacol Biochem Behav. 2003 Sep;76(2):351-60. doi: 10.1016/j.pbb.2003.08.008. PMID 14592688
- [Background] Spring B, Pingitore R, McChargue DE. Reward value of cigarette smoking for comparably heavy smoking schizophrenic, depressed, and nonpatient smokers. Am J Psychiatry. 2003 Feb;160(2):316-22. doi: 10.1176/appi.ajp.160.2.316. PMID 12562579
- [Background] Johnsen L, MacKirnan D, Spring B, Pingitore R, Sommerfeld BK. Smoking as subculture? Influence on Hispanic and non-Hispanic White women's attitudes toward smoking and obesity. Health Psychol. 2002 May;21(3):279-87. doi: 10.1037//0278-6133.21.3.279. PMID 12027034
- [Background] Richmond M, Spring B, Sommerfeld BK, MeChargue D. Rumination and cigarette smoking: a bad combination for depressive outcomes? J Consult Clin Psychol. 2001 Oct;69(5):836-40. doi: 10.1037//0022-006x.69.5.836. PMID 11680561
- [Background] Borrelli B, Spring B, Niaura R, Kristeller J, Ockene JK, Keuthen NJ. Weight suppression and weight rebound in ex-smokers treated with fluoxetine. J Consult Clin Psychol. 1999 Feb;67(1):124-31. doi: 10.1037//0022-006x.67.1.124. PMID 10028216
- [Derived] Schneider KL, Hedeker D, Bailey KC, Cook JW, Spring B. A comment on analyzing addictive behaviors over time. Nicotine Tob Res. 2010 Apr;12(4):445-8. doi: 10.1093/ntr/ntp213. Epub 2010 Jan 25. PMID 20100810